CLINICAL TRIAL: NCT01444092
Title: A Multicenter, Open Label, Non-comparative Study to Evaluate the Safety of Entocort EC for the Treatment of Crohn's Disease in Paediatric Subjects Aged 5 to 17 Years, Inclusive
Brief Title: Safety Study of Entocort for Children With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9422C00001
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Budesonide

ARMS (1):
- Entocort (Experimental): Study Medication
  Interventions: Drug: Entocort

INTERVENTIONS:
Drug: Entocort — Entocort capsules, oral

SUMMARY:
A Safety Study using Entocort EC for children with mild to moderate Crohn's Disease

DETAILED DESCRIPTION:
A Multicenter, Open label, Non-comparative Study to Evaluate the Safety of Entocort EC for the Treatment of Crohn's Disease in Paediatric Subjects Aged 5 to 17 Years, Inclusive

ELIGIBILITY:
Inclusion Criteria:

* All male and female subjects must be aged 5 to 17, inclusive, and must not have reached their 18th birthday by the estimated final office visit.
* Subject must be diagnosed with active Crohn's disease of the ileum and/or ascending colon confirmed by endoscopic and/or radiographic evidence, and/or evidence of mucosal erosions and/or histology.
* Subjects with mild to moderate Crohn's disease.
* All subjects must have a stool analysis negative for Clostridium difficile toxin, Yersinia enterolytica, Campylobacter jejuni, Salmonella, Shigella, within the 30 days prior to visit 1.
* All subjects must have had laboratory assessments within 7 days prior to visit 1.
* All subjects must weigh >= 15 kg at time of enrollment

Exclusion Criteria:

* Subjects who have had any previous intestinal resection proximal to and including the ascending colon
* Subjects with evidence of severe active Crohn's disease and/or, stricturing and prestenotic dilatation, clinical evidence of obstruction, perirectal abscess, perirectal disease with active draining fistulas, perforation, or any septic complications
* Subjects who do not have a negative stool analysis, within the 30 days prior to visit 1
* Subjects who have been screened/or enrolled in this study previously within the last 30 days
* Subjects with morning cortisol level <150 nmol/l (5.4 ug/dl) or DHEA-S below normal range for age and gender

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Cohen, MD, Principal Investigator — Children's Center for Digestive Healthcare, LLC, Atlanta, Georgia, USA and Emory University School of Medicine, Atlanta, Georgia, USA; Stefan Eklund, MD, Study Director — AstraZeneca Pharmaceuticals, Mölndal, Sweden
Locations (24):
- United States (11):
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Saint Paul, Minnesota
  - Research Site, Mays Landing, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Nashville, Tennessee
- Canada (3):
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
- Research Site, München, Germany
- Italy (4):
  - Research Site, Florence
  - Research Site, Messina
  - Research Site, Napoli
  - Research Site, Roma
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw

REFERENCES:
- [Derived] Cohen SA, Aloi M, Arumugam R, Baker R, Bax K, Kierkus J, Koletzko S, Lionetti P, Persson T, Eklund S. Enteric-coated budesonide for the induction and maintenance of remission of Crohn's disease in children. Curr Med Res Opin. 2017 Jul;33(7):1261-1268. doi: 10.1080/03007995.2017.1313213. Epub 2017 Apr 19. PMID 28420280
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=648&filename=D9422C00001_Clinical_Trial_Disclosure_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 patients were screened/enrolled, but only 108 received treatment. The other 15 did not meet the inclusion/exclusion criteria. They only appear in the disposition tables in the CSR (Tables 8 and 10) and did not "start" in the study.
Pre-assignment Details: 123 patients were screened/enrolled, but only 108 received treatment. The other 15 did not meet the inclusion/exclusion criteria. They only appear in the disposition tables in the CSR (Tables 8 and 10) and did not "start" in the study.
Groups:
- Entocort: Entocort™ EC 9/6/3 mg
Period: Overall Study
Arm/Group | Entocort
Started | 108
INFORMED CONSENT OBTAINED | 108
Completed | 91
Not Completed | 17
Not completed — Adverse Event | 8
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other Eligibility criteria | 7

BASELINE CHARACTERISTICS:
Arm/Group | Entocort
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 13.7 (2.41) [6 to 17]
Age, Customized [Number; unit: Participants]
  =<8 Yrs | 5
  >8 Yrs | 103
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 57
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1
  Black Or African American | 4
  Other | 3
  White | 100

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event
Description: Number of patients with at least one adverse event
Time Frame: 12 weeks
Population: Safety analysis set
Measure: Number; unit: Patients
Arm/Group | Entocort
Number analyzed (Participants) | 108
Patients | 79

2. Secondary Outcome: PCDAI
Description: Paediatric Crohn's Disease Activity Index. Range from 0 (best) to 100 (worst).
Time Frame: Baseline to 8 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Entocort
Number analyzed (Participants) | 105
Units on a scale
  Baseline (Day1) | 19.10 (10.1)
  Change after 8 weeks | -10.0 (10.1)

3. Secondary Outcome: IMPACT 3
Description: IMPACT 3 is a self-administered QoL form. The score ranges from 35 (poor) to 175 (best).
Time Frame: Baseline to 8 weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Entocort
Number analyzed (Participants) | 107
Units on a scale
  Baseline (Day 1) | 132.1 (18.8)
  Change after 8 weeks | 7.8 (13.3)

ADVERSE EVENTS:
Arm/Group | Entocort
Serious Adverse Events (participants affected / at risk) | 8/108
Other Adverse Events (participants affected / at risk) | 78/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entocort (N=108)
Crohn's disease (Gastrointestinal disorders) | 4 (4)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entocort (N=108)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Cushingoid (Endocrine disorders) | 13 (13)
Iritis (Eye disorders) | 1 (1)
Scleritis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 16 (16)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 2 (2)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1)
Anal skin tags (Gastrointestinal disorders) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1)
Cheilosis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 6 (6)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chest pain (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Tenderness (General disorders) | 1 (1)
Acarodermatitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4)
Otitis externa (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (4)
Rectal abscess (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1)
Blood cortisol decreased (Investigations) | 1 (1)
Blood cortisol increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Mean cell volume decreased (Investigations) | 1 (1)
Occult blood positive (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 3 (3)
Urine output decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 17 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (9)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 6 (6)
Irritability (Psychiatric disorders) | 14 (14)
Mood swings (Psychiatric disorders) | 3 (3)
Sleep disorder (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menstrual disorder (Reproductive system and breast disorders) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 15 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 (2)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Hirsutism (Skin and subcutaneous tissue disorders) | 5 (5)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin striae (Skin and subcutaneous tissue disorders) | 2 (2)
Pallor (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No